CLINICAL TRIAL: NCT05932212
Title: A Multicenter, Open-label, Phase II Study of AK104 in the Treatment of Recurrent or Metastatic Vulvar Cancer
Brief Title: AK104 for Recurrent or Metastatic Vulvar Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK104-218
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Vulvar Cancer
Keywords: PD-1/CTLA-4; vulvar cancer
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: AK104 (Experimental): AK104 monotherapy
  Interventions: Drug: AK104
- Cohort B: AK104+chemotherapy (Experimental): AK104 combined with platinum-based chemotherapy (paclitaxel+ cisplatin or carboplatin)
  Interventions: Drug: AK104+ Paclitaxel+Cisplatin or Carboplatin

INTERVENTIONS:
Drug: AK104 — AK104 15mg/kg intravenously(IV) every 3 weeks (Q3W), until progressive disease, unacceptable toxicity, completion of 2 years treatment or withdrawal of consent.
  Other Names: Cadonilimab
  Arms: Cohort A: AK104
Drug: AK104+ Paclitaxel+Cisplatin or Carboplatin — AK104 (10 mg/kg) + paclitaxel (175 mg/m2)+ cisplatin (50 mg/m2) or carboplatin (AUC 4-5) , IV, Q3W, for up to 6 cycles, followed by maintenance therapy of AK104 10 mg/kg Q3W until disease progression, intolerable toxicity, withdrawal of consent, or completion of 2 years treatment.
  Arms: Cohort B: AK104+chemotherapy

SUMMARY:
This is a multicenter, open-label, phase II clinical study, aiming to the evaluate the efficacy and safety of AK104 (an anti- PD-1 and CTLA-4 bispecific antibody), alone or combined with chemotherapy, in subjects with recurrent or metastatic vulvar cancer not amenable to curative surgery or radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

Age >=18 and <=80. ECOG of 0 or 2. Life expectancy ≥ 3 months. Histologically confirmed vulvar cancer (squamous cell carcinoma or adenosquamous carcinoma), not amenable to curative surgery or radical radiotherapy.

For Cohort A, subjects should have experienced failure on at least one previous systemic therapy, or intolerance to standard therapy.

At least one measurable tumor lesion per RECIST v1.1. Adequate organ function as assessed in the laboratory tests. Female subjects of childbearing potential must have a negative serum pregnancy test prior to the the first administration and agree to use effective methods of contraception

Exclusion Criteria:

Subjects with other histopathological types of vulvar cancer, such as melanoma, sarcoma, etc.

Systemic or curative (surgery or radiotherapy) anti-tumor therapy within 4 weeks prior to the first administration.

Previous treatment with immune checkpoint inhibitors (e.g., anti-PD-1 antibody, anti-PD-L1 antibody, anti-CTLA-4 antibody, etc.).

Active or potentially recurrent autoimmune disease.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) assessed by investigator. | Up to approximately 1 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR per RECIST v1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) Assessed by investigator | Up to approximately 2 years
  The time from the first administration to the first documented progressive disease (PD) or death due to any cause, whichever occurs first
Duration of Response (DOR) Assessed by investigator | Up to approximately 2 years
  Measured from the date of partial or complete response to therapy until the disease progression per RECIST v1.1 criteria
Disease control rate (DCR) Assessed by investigator | Up to approximately 1 years
  The proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥6 weeks) based on RECIST
Time to Response (TTR) Assessed by investigator | Up to approximately 1 years
  The time from the first administration to the date of documented CR or PR
Overall survival (OS) | Up to approximately 2 years
  The time from the first administration to death due to any cause
Adverse Events (AEs) | Up to approximately 2 years
  Characterization of incidence, severity and abnormal clinically significant manifestation or laboratory findings.
serum concentrations of AK104 | Up to approximately 2 years
  assessment of PK include serum concentrations of AK104 at different timepoints after study drug administration
Antidrug antibodies (ADA) of AK104 | Up to approximately 2 years
  Proportion of subjects who develop detectable anti-drug antibodies (ADAs)

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Clinical oncology school of Fujian Medical University, Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yant-Sen Memorial Hospital, Guangzhou, Guangdong
  - The Fourth Hospital of Hebei Medical University, Shijiangzhuang, Hebei
  - Liaoning Cancer Hospital & Insitut, Shenyang, Liaoning
  - Tianjin medical university Cancer Institut & Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No